CLINICAL TRIAL: NCT00248937
Title: A Pilot Study of Changing Medication Adherence In Hypertensive African-American Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Mary E. Charlson, MD, Weill Medical College
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: N01-HC-25196 (0203-703); N01HC25196 (NIH)
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-04

CONDITIONS: Hypertension
Keywords: African-American; Hypertension; Medication adherence; Risk reduction
MeSH Terms: conditions — Hypertension; Medication Adherence; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Positive affect and self-affect induction

SUMMARY:
We will conduct an empirical test of the two intervention approaches under study. Specifically, we seek to determine the potential differential impact of positive affect induction and self affirmation.

DETAILED DESCRIPTION:
We are interested in achieving an empirical test of the two intervention approaches under study. Specifically, we seek to determine the potential differential impact of positive affect induction and self affirmation following the qualitative phase.

1. Positive affect induction: We will tests two types of positive affect induction. 1) sending patients a small gift, and 2) reminding patients of positive thoughts about themselves.

   Gift: Prior to a telephone call, patients in the positive affect condition will receive a small gift.

   Positive thoughts about themselves: Patients will be asked to describe a time when someone was helpful to them, and they felt good about it , and were nice to them in return.
2. Self affirmation: consists of a series of items reminding people of their core values.
3. Control: Control patients will have neither self affirmation nor gifts.

Follow-up: At two weeks after enrollment all patients will be called to ascertain impact of the pilot intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be self-identified as African-Americans.
2. All patients must be aged 18 years and older.
3. All patients must be diagnosed as having hypertension: For this project, hypertension will be defined according to the widely accepted criteria of the 6th Joint National Committee (JNC VI) Guidelines on Prevention, Detection, Evaluation and Treatment of Hypertension, which is a systolic blood pressure > 140 mm hg or a diastolic blood pressure > 90 mm hg or if participants are taking any prescribed antihypertensive medication.
4. Patients must be able to provide informed consent in English.

Exclusion Criteria:

1. Patients who are unable to walk several blocks for any reason.
2. Patients who refused to participate
3. Patients who are unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-02; Study Completion 2004-06

PRIMARY OUTCOMES:
Within patient change on the Positive and Negative Affect Scale

CONTACTS AND LOCATIONS:
Overall Officials: Carla Boutin-Foster, MD, MS, Principal Investigator — Weill Medical College of Cornell University; Gbenga Ogedegbe, MD, MS, Principal Investigator — Columbia University; Mary E Charlson, MD, Study Director — Weill Medical College of Cornell University
Locations (1):
- The New York Presbyterian Hospital-Weill Medical Center, New York, New York, United States